CLINICAL TRIAL: NCT04626414
Title: A Randomized, Open-Label, Single Dose, Four-Way Crossover, Phase I Study to Compare the Pharmacokinetics of Ferric Maltol Capsules and Oral Suspension Under Fasted and Fed Conditions in Adult Healthy Volunteers
Brief Title: Four-Way Crossover Study to Compare Ferric Maltol Capsules and Oral Suspension in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shield Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ST10-01-104
Record Dates: First submitted 2020-10-22; First posted 2020-11-12 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Anemia, Iron Deficiency
Keywords: iron deficiency, anaemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric maltol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1:1:1 to one of the treatment sequences. ie. single dose of 30 mg ferric maltol capsule in a fed condition single dose of 30 mg (5 ml) ferric maltol suspension in a fed condition single dose of 30 mg ferric maltol capsule in a fasted condition single dose of 30 mg (5 ml) ferric maltol suspension in a fasted condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 30 mg ferric maltol capsule in a fed condition (Active Comparator): Single dose of 30 mg ferric maltol capsule in a fed condition
  Interventions: Drug: Ferric maltol capsule
- 30 mg ferric maltol capsule in a fasted condition (Active Comparator): Single dose of 30 mg ferric maltol capsule in a fasted condition
  Interventions: Drug: Ferric maltol capsule
- 30 mg (5 ml) ferric maltol suspension in a fed condition (Experimental): Single dose of 30 mg (5 ml) ferric maltol suspension in a fed condition
  Interventions: Drug: Ferric maltol suspension
- 30 mg (5 ml) ferric maltol suspension in a fasted condition (Experimental): Single dose of 30 mg (5 ml) ferric maltol suspension in a fasted condition
  Interventions: Drug: Ferric maltol suspension

INTERVENTIONS:
Drug: Ferric maltol capsule — single dose of 30 mg capsule
  Other Names: ST10, Feraccru; Accrufer
  Arms: 30 mg ferric maltol capsule in a fasted condition; 30 mg ferric maltol capsule in a fed condition
Drug: Ferric maltol suspension — single dose of 30mg (5ml) oral suspension
  Other Names: ST10
  Arms: 30 mg (5 ml) ferric maltol suspension in a fasted condition; 30 mg (5 ml) ferric maltol suspension in a fed condition

SUMMARY:
The purpose of the study is to compare the Pharmacokinetics (PK) of the new ferric maltol suspension, in adults, with the existing ferric maltol capsule.

DETAILED DESCRIPTION:
Open-label, Phase 1, four way crossover study to compare the PK of the new ferric maltol suspension, in healthy volunteers, with the existing ferric maltol capsules under fed and fasted conditions.

32 subjects will be randomised to 1:1:1:1 ratio to receive one of the treatment sequences.

Based on the randomised sequence, subjects will receive a single dose of 30mg ferric maltol capsule in a fed/ fasted condition and 30 mg (5ml) ferric maltol suspension in a fed/ fasted condition.

Subject participation in the study will consist of 3 periods:

1. Screening: up to 14 days
2. Randomised treatment: 8 days
3. Post-treatment follow up: 3-7 days following drug discontinuation

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met for a subject to participate in the study:

1. Must voluntarily sign and date each Institutional Review Board (IRB)-approved informed consent form (ICF) prior to the initiation of any screening or study-specific procedures.
2. Willing and able to comply with study requirements.
3. Healthy adult subjects 18 to 55 years of age, inclusive at the time of informed consent.
4. Body Mass Index (BMI) of 18-32 kg/m2 inclusive
5. Female subjects of childbearing potential must not be planning a pregnancy or be pregnant or lactating. All female subjects must have a negative result for the pregnancy tests performed at screening and each treatment period.
6. Female subjects of childbearing potential (including perimenopausal females who have had a menstrual period within 1 year prior to screening) must agree to use a reliable method of contraception until study completion and for at least 4 weeks following their final study visit. Reliable contraception is defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as hormonal contraception (oral, implants, injection, ring, or patch) and intrauterine contraceptive devices (IUDs), at least 3 months prior to Screening, or a vasectomized partner.

   Note: complete abstinence from sexual intercourse is an acceptable form of contraceptive practice.
7. Female subjects of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral, tubal ligation, bilateral salpingectomy, and/or bilateral oophorectomy at least 26 weeks before the Screening Visit) or post-menopausal, defined as spontaneous amenorrhea for at least 2 years
8. Male subjects with partners of childbearing potential must have had surgical sterilization (vasectomy) at least 26 weeks prior to Screening or use a male barrier method of contraception (i.e. male condom with spermicide) during any sexual intercourse from Study Day -1 (beginning of confinement) until 3 months after the Follow-up Visit.

   Note: Complete abstinence from sexual intercourse is an acceptable form of contraceptive practice.
9. Male subjects must agree to abstain from sperm donation from initial study drug administration through 3 months after administration of the last dose of study drug.

Exclusion Criteria:

A subject who meets any of the following criteria is not eligible for participation in the study.

1. Known hypersensitivity or allergy to the active substance or excipients of Ferric maltol oral suspension or capsules;
2. Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurological, or psychiatric disease, as determined by the Investigator;
3. Presence or history of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines;
4. Recent (within 6 months of screening) history of drug or alcohol abuse;
5. Positive screen results for drugs of abuse, alcohol at screening or Study Day -1 of Period1;
6. Consumption of alcohol within 72 hrs prior to study drug administration;
7. Positive test result for hepatitis B surface antigen (HBSaAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening;
8. Donation or loss of 550 mL or more blood volume or receipt of a transfusions of any blood product within 8 weeks prior to study drug administration and 14 days for plasma donation unless medically inadvisable;
9. Use of any over the counter medications, including herbal product within 7 days prior to Screening until study completion. Except for ordinary pain (e.g. headache), some analgesics (mainly paracetamol) and contraception which have no drug interactions with the study products may be given;
10. Has received within 28 days prior to Screening intramuscular or intravenous (IV) injection or administration of depot iron preparation;
11. Has received oral iron supplementation within 7 days prior to Screening;
12. Has concomitant disease that would significantly compromise iron absorption or absorbed iron utilization such as swallowing disorders, gastric pH-disturbance and/or extensive small bowel resection;
13. Scheduled or expected hospitalization and/or surgery during the course of the study;
14. Diagnosed to be COVID-19 positive by polymerase chain reaction testing (SARS-CoV-2-RTPCR positive) of a respiratory specimen (preferably a nasopharyngeal swab) on Day -2;
15. Participation in any other interventional clinical study within 28 days prior to Screening;
16. Any other unspecified reason that, in the opinion of the Investigator or the Sponsor makes the subject unsuitable for enrolment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Mitchell, DPhil, Study Director — Shield Therapeutics
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 subjects recruited. 8 subjects randomised to each sequence.
Groups:
- Ferric Maltol Sequence A: Period 1 capsule-fed; Period 2 suspension-fed; Period 3 capsule-fasted; Period 4 suspension-fasted.
- Ferric Maltol Sequence B: Period 1 suspension-fasted; Period 2 capsule-fed; Period 3 suspension-fed; Period 4 capsule-fasted.
- Ferric Maltol Sequence C: Period 1 capsule-fasted; Period 2 suspension-fasted; Period 3 capsule-fed; Period 4 suspension-fed.
- Ferric Maltol Sequence D: Period 1 suspension-fed; Period 2 capsule-fasted; Period 3 suspension-fasted; Period 4 capsule-fed.
Period: Overall Study
Arm/Group | Ferric Maltol Sequence A | Ferric Maltol Sequence B | Ferric Maltol Sequence C | Ferric Maltol Sequence D
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall demographic and baseline characteristics of the randomised population. The Randomized population is defined as all subjects who are randomized. The FAS is defined as all subjects who have had at least one dose of study drug and who have at least one evaluable post-dose PK sample.
Groups:
- Ferric Maltol Sequence A: Period 1 capsule-fed; Period 2 suspension fed; Period 3 capsule fasted; Period 4 suspension fasted.
- Ferric Maltol Sequence B: Period 1 suspension fasted; Period 2 capsule-fed; Period 3 suspension fed; Period 4 capsule fasted.
- Ferric Maltol Sequence C: Period 1 capsule fasted; Period 2 suspension fasted; Period 3 capsule fed; Period 4 suspension fed.
- Ferric Maltol Sequence D: Period 1 suspension fed; Period 2 capsule fasted; Period 3 suspension fasted; Period 4 capsule fed.
- Total: Total of all reporting groups
Arm/Group | Ferric Maltol Sequence A | Ferric Maltol Sequence B | Ferric Maltol Sequence C | Ferric Maltol Sequence D | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (9.33) | 34.00 (11.05) | 33.6 (6.44) | 40.5 (8.82) | 36.18 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 5 | 15
  Male | 5 | 5 | 4 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 8 | 8 | 7 | 6 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 6 | 5 | 5 | 24
  White | 0 | 2 | 3 | 3 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Maximum Serum Concentration (Cmax) of Total Iron in Fasted Condition
Description: Ratio of maximum serum concentration (Cmax) of total iron in combined periods of fasted condition between ferric maltol capsule and ferric maltol suspension.
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose in combined fasted condition
Population: Full Analysis Set Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- Ferric Maltol Capsule and Ferric Maltol Suspension in a Fasted Condition: 30 mg ferric maltol capsule and 30 mg (5 ml) ferric maltol suspension in a fasted condition
Arm/Group | Ferric Maltol Capsule and Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32
ratio | 69.94 [61.75 to 79.23]

2. Primary Outcome: Ratio of Maximum Serum Concentration (Cmax) of Total Iron in Combined Periods of Fed Condition
Description: Ratio of maximum serum concentration (Cmax) of total iron in combined periods of fed condition between ferric maltol capsule and ferric maltol suspension
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose in combined fed condition
Population: Full analysis set population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- Ferric Maltol Capsule Fed and Ferric Maltol Suspension Fed: 30 mg ferric maltol capsule and 30 mg (5 ml) ferric maltol suspension in a fed condition
Arm/Group | Ferric Maltol Capsule Fed and Ferric Maltol Suspension Fed
Number analyzed (Participants) | 32
ratio | 99.11 [87.50 to 112.27]

3. Primary Outcome: Ratio of Area Under the Curve (AUClast) of Total Serum Iron in Combined Period of Fasted Condition
Description: Ratio of area under the curve (AUClast) of total serum iron in combined periods of fasted condition between ferric maltol capsule and ferric maltol suspension
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose in combined fasted condition
Population: FAS
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- Ferric Maltol Capsule Fasted and Ferric Maltol Suspension Fasted: 30 mg ferric maltol capsule and 30 mg (5 ml) ferric maltol suspension in a fasted condition
Arm/Group | Ferric Maltol Capsule Fasted and Ferric Maltol Suspension Fasted
Number analyzed (Participants) | 32
ratio | 77.54 [70.38 to 85.42]

4. Primary Outcome: Ratio of Area Under the Curve (AUClast) of Total Serum Iron in Combined Period of Fed Condition
Description: Ratio of area under the curve (AUClast) of total serum iron in combined periods of fed condition between ferric maltol capsule and ferric maltol suspension
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose in combined fed condition
Population: Full analysis set population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Ferric Maltol Capsule Fed and Ferric Maltol Suspension Fed
Number analyzed (Participants) | 32
ratio | 96.99 [88.04 to 106.86]

5. Primary Outcome: Ratio of Maximum Serum Concentration (Cmax) of Total Iron in Fasted vs Fed Condition in Ferric Maltol Capsule
Description: Ratio of maximum serum concentration (Cmax) of total iron in fasted vs fed condition in 30mg ferric maltol capsule
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose on both PK days
Population: Full Analysis Set Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- Ferric Maltol Capsule in Fed vs. Fasted Condition: 30 mg ferric maltol capsule in fed vs fasted condition
Arm/Group | Ferric Maltol Capsule in Fed vs. Fasted Condition
Number analyzed (Participants) | 32
ratio | 147.27 [130.01 to 166.81]

6. Primary Outcome: Ratio of Area Under the Curve (AUClast) of Total Serum Iron in Fasted vs. Fed Condition in Ferric Maltol Capsule
Description: Ratio of area under the curve (AUClast) of total serum iron in fasted vs fed condition in 30 mg ferric maltol capsule
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose in both PK days
Population: FAS
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Ferric Maltol Capsule in Fed vs. Fasted Condition
Number analyzed (Participants) | 32
ratio | 134.25 [121.86 to 147.91]

7. Primary Outcome: Ratio of Maximum Serum Concentration (Cmax) of Total Iron in Fasted vs Fed Condition in Ferric Maltol Suspension
Description: Ratio of maximum serum concentration (Cmax) of total iron in fasted vs fed condition in 30mg (5ml) ferric maltol suspension
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose on both PK days
Population: FAS
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- Ferric Maltol Suspension in Fed vs Fasted Condition: 30mg (5ml) ferric maltol suspension in fed vs fasted condition
Arm/Group | Ferric Maltol Suspension in Fed vs Fasted Condition
Number analyzed (Participants) | 32
ratio | 103.93 [91.75 to 117.72]

8. Primary Outcome: Ratio of Area Under the Curve (AUClast) of Total Serum Iron in Fasted vs. Fed Condition in Ferric Maltol Suspension
Description: Ratio of area under the curve (AUClast) of total serum iron in fasted vs fed condition in 30mg (5ml) ferric maltol suspension
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose in both PK days
Population: FAS
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- Ferric Maltol Suspension in Fasted vs Fed Condition: 30mg (5ml) ferric maltol suspension in fasted vs fed condition
Arm/Group | Ferric Maltol Suspension in Fasted vs Fed Condition
Number analyzed (Participants) | 32
ratio | 107.32 [97.41 to 118.24]

9. Secondary Outcome: PK Analysis of Total Serum Iron Concentration; AUCinf in Fasted and Fed Conditions
Description: Descriptive statistics of total serum iron concentration; Area Under the Curve (AUCinf) by formulation (suspension or capsule) and condition (fed and fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS - If the Lambda z was not assigned, the values of associated PK parameters AUCinf was not calculated
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 10 | 19 | 10 | 13
h*ng/mL | 2922.46 (1052.46) | 3694.05 (1561.138) | 3330.98 (2128.861) | 3445.41 (2615.954)

10. Secondary Outcome: PK Analysis of Baseline Corrected Serum Iron Concentration; Cmax in Fasted and Fed Conditions
Description: Descriptive statistics of baseline corrected serum iron concentration; Maximum Concentration (Cmax), by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng/mL | 44.469 (73.0572) | 89.938 (50.9927) | 40.219 (52.9715) | 33.250 (23.0637)

11. Secondary Outcome: PK Analysis of Baseline Corrected Serum Iron Concentration; AUClast in Fasted and Fed Conditions
Description: Descriptive statistics of baseline corrected serum iron concentration; area under the Curve from pre-dose to last measurable concentration by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
h*ng/mL | 56.150 (964.9572) | 691.392 (791.8671) | 2.503 (889.0745) | -9.436 (693.2830)

12. Secondary Outcome: PK Analysis of Baseline Corrected Serum Iron Concentration; AUCinf in Fasted and Fed Conditions
Description: Descriptive statistics of baseline corrected serum iron concentration; Area Under the Curve from 0-infinity by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS. If the Lambda z was not assigned, the values of associated PK parameters AUCinf was not calculated.
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: PK Analysis of Maltol Glucuronide; Cmax in Fasted and Fed Conditions
Description: Descriptive statistics of Maximum plasma Concentration (Cmax) of plasma maltol glucuronide by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng/mL | 3579.063 (1668.2120) | 5126.250 (1996.0748) | 3597.500 (1776.4390) | 7685.0 (1920.3797)

14. Secondary Outcome: PK Analysis of Maltol Glucuronide; AUClast in Fasted and Fed Conditions
Description: Descriptive statistics of maltol glucuronide; Area Under the Curve from pre-dose to last measurable concentration by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
h*ng/mL | 7335.93 (2449.530) | 9083.82 (2902.863) | 7802.52 (2585.848) | 10410.89 (2631.072)

15. Secondary Outcome: PK Analysis of Maltol; Cmax in Fasted and Fed Conditions
Description: Descriptive statistics of Maximum plasma Concentration (Cmax) of plasma maltol by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng/mL | 16.994 (18.5420) | 20.531 (16.0714) | 33.600 (37.0501) | 34.656 (25.2179)

16. Secondary Outcome: PK Analysis of Maltol; AUClast in Fasted and Fed Conditions
Description: Descriptive statistics of maltol; Area Under the Curve from pre-dose to last measurable concentration by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS - If the Lambda z was not assigned, the values of associated PK parameters AUC last was not calculated.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 20 | 27 | 28 | 31
h*ng/mL | 28.61 (21.924) | 17.29 (15.274) | 39.13 (44.525) | 22.41 (16.879)

17. Secondary Outcome: PK Analysis of TSAT; Cmax in Fasted and Fed Conditions
Description: Descriptive statistics of Maximum Concentration (Cmax) of transferrin saturation by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng/mL | 32.750 (18.4793) | 43.031 (12.9428) | 30.344 (12.5970) | 30.188 (9.3892)

18. Secondary Outcome: PK Analysis of TSAT; AUClast in Fasted and Fed Conditions
Description: Descriptive statistics of transferrin saturation; Area Under the Curve from pre-dose to last measurable concentration by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
h*ng/mL | 509.90 (201.915) | 644.62 (176.724) | 484.64 (153.990) | 513.62 (193.642)

19. Secondary Outcome: PK Analysis of TIBC; Cmax in Fasted and Fed Conditions
Description: Descriptive statistics of Maximum Concentration (Cmax) of Total Iron Binding Capacity (TIBC) by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng/mL | 393.688 (50.5208) | 394.781 (50.9913) | 396.938 (73.3577) | 394.656 (46.5310)

20. Secondary Outcome: PK Analysis of TIBC; AUClast in Fasted and Fed Conditions
Description: Descriptive statistics of Total Iron Binding Capacity (TIBC); Area Under the Curve from pre-dose to last measurable concentration by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
h*ng/mL | 8719.09 (1097.981) | 8880.52 (1165.547) | 8718.02 (1195.335) | 8878.43 (1069.977)

21. Secondary Outcome: Summary of Serious Adverse Events
Description: Descriptive statistics of Serious Adverse Events by formulation (suspension or capsule) and condition (fed and fasted)
Time Frame: up to 2 weeks following last dose
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: PK Analysis of UIBC; Cmax in Fasted and Fed Conditions
Description: Descriptive statistics of Maximum Concentration (Cmax) of Unsaturated Iron Binding Capacity (UIBC) by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng/mL | 329.750 (57.3298) | 323.250 (59.0172) | 331.250 (82.0668) | 322.375 (55.7018)

23. Secondary Outcome: PK Analysis of UIBC; AUClast in Fasted and Fed Conditions
Description: Descriptive statistics of Unsaturated Iron Binding Capacity (TIBC); Area Under the Curve from pre-dose to last measurable concentration by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1,1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
h*ng/mL | 6836.84 (1303.757) | 6432.85 (1052.589) | 6939.53 (1159.295) | 6978.71 (1182.131)

24. Secondary Outcome: PK Analysis of Transferrin; Cmax in Fasted and Fed Conditions
Description: Descriptive statistics of transferrin; Maximum concentration (Cmax) from pre-dose to last measurable concentration by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng/mL | 304.063 (42.7332) | 302.594 (44.5051) | 300.688 (42.3316) | 303.031 (40.1670)

25. Secondary Outcome: PK Analysis of Transferrin; AUClast in Fasted and Fed Conditions
Description: Descriptive statistics of transferrin; Area Under the Curve from pre-dose to last measurable concentration by formulation (suspension or capsule) and condition (fed or fasted)
Time Frame: Pre-dose and 0.15, 0.30, 0.45, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose
Population: FAS
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
h*ng/mL | 6711.95 (965.632) | 6774.38 (948.865) | 6701.92 (980.522) | 6837.00 (936.103)

26. Secondary Outcome: Treatment-Emergent Adverse Events
Description: Treatment-Emergent Adverse Events from Day 1 to Day 22 (Study completion)
Time Frame: From first dose of ferric maltol on Day 1 to study completion
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 0 | 2 | 3 | 3

27. Secondary Outcome: TEAE Leading to Premature Discontinuation of Study Drug/PK Assessments
Description: TEAE leading to premature discontinuation of study drug/PK assessments from Day 1 to study completion
Time Frame: From first dose of ferric maltol on Day 1 to study completion
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

28. Secondary Outcome: Vital Signs - Blood Pressure, Change From Day 1 to Day 8
Description: Descriptive statistics for changes in blood pressure from Screening to Day 8
Time Frame: Screening to Day 8
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Sequence A: Period 1 capsule-fed; Period 2 suspension-fed; Period 3 capsule-fasted; Period 4 suspension-fasted
- Sequence B: Period 1 suspension-fasted; Period 2 capsule-fed; Period 3 suspension-fed; Period 4 capsule-fasted
- Sequence C: Period 1 capsule-fasted; Period 2 suspension-fasted; Period 3 capsule-fed; Period 4 suspension-fed
- Sequence D: Period 1 suspension-fed; Period 2 capsule-fasted; Period 3 suspension-fasted; Period 4 capsule-fed
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Number analyzed (Participants) | 8 | 8 | 8 | 8
mmHg
  Diastolic blood pressure | -0.5 (3.02) | -0.3 (6.71) | -3.6 (7.58) | -2.4 (4.63)
  Systolic blood pressure | -3.6 (6.25) | -4.6 (10.90) | -4.9 (14.59) | -0.1 (7.16)

29. Secondary Outcome: Vital Signs - Heart Rate, Change From Day 1 to Day 7
Description: Descriptive statistics for changes in heart rate from Screening to Day 7
Time Frame: Screening to Day 7
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Number analyzed (Participants) | 8 | 8 | 8 | 8
beats/min | -0.8 (10.26) | 8.1 (8.69) | 11.1 (11.23) | 3.1 (6.13)

30. Secondary Outcome: Summary of Received Concomitant Medication by Formulation
Description: Number of participants having received concomitant medications by formulation (suspension or capsule)
Time Frame: Day 1 to Day 8 (24 hrs post-dose of last dosing)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
Number analyzed (Participants) | 32 | 32 | 32 | 32
participants | 2 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: 8 days
Arm/Group | 30 mg Ferric Maltol Capsule in a Fed Condition | 30 mg Ferric Maltol Capsule in a Fasted Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 2/32 | 3/32 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg Ferric Maltol Capsule in a Fed Condition (N=32) | 30 mg Ferric Maltol Capsule in a Fasted Condition (N=32) | 30 mg (5 ml) Ferric Maltol Suspension in a Fed Condition (N=32) | 30 mg (5 ml) Ferric Maltol Suspension in a Fasted Condition (N=32)
Vessel puncture site pain (General disorders) | 0 | 1 (1) | 1 (1) | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0
Headache (Nervous system disorders) | 0 | 1 (1) | 0 | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04626414/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04626414/SAP_001.pdf